CLINICAL TRIAL: NCT00976586
Title: In Vitro Observation of Chromosome Recombination and Treatment in Vitro
Brief Title: Role of Pseudogene in Incontinentia Pigmenti, and Its Potential Treatment
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, National Taiwan University Hospital, Attending, National Taiwan University Hospital
Other Study IDs: 200812061R
Record Dates: First submitted 2009-09-10; First posted 2009-09-14 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Incontinentia Pigmenti
Keywords: Incontinentia pigmenti; recombination; IKBKG; IKBKGP
MeSH Terms: conditions — Incontinentia Pigmenti

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood for DNA and plasma. Skin for cultured fibroblast
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients wiht Incontinentia Pigmenti: Patients wiht Incontinentia Pigmenti

SUMMARY:
Incontinentia Pigmenti (IP) is an X-linked dominant ectodermal dysplastic disorder. It is due to loss of function of NF-Kappa B Essential Modulator (NEMO, inhibitor of Kappa light polypeptide gene enhancer in B cells, Kinase of Gamma, IKBKG), an important regulator of the NF-kB pathway. Major clinical manifestations of IP include swirling skin pigmentary changes, and anomalies in organs including the eyes, dental, bones, nervous system, and heart. Affected male mostly die before birth. Older patients might have immunodeficiency, psychomotor retardation, and seizures. Prenatal diagnosis is difficult. IKBKG gene is 35 kb in length, and contains 10 exons. A pseudogene (∆NEMO, IKBKGP), located distal and in inverse direction to the true gene, contains only exon 3-10. In patients with IP, the most common mutation was exon 4-10 large deletion. But the investigators have found small mutations derived from the pseudogene in Taiwanese patients.

The three aims of this study are the role of pseudogene in IP, the frequency of recombination between IKBKG and IKBKGP, and possible treatment. To achieve the first aim, the investigators first develop a pseudogene-specific polymerase chain reaction (PCR). The investigators will first obtain the frequency of IKBKGP gene mutation in normal individuals. The investigators will then detect IKBKGP related mutations in IP patients presenting classical or non-classical symptoms. The latter group of patients, who may have isolated hair, teeth, retinal, or immune problems, are more likely to be caused by point mutations. The second aim of this study is to estimate the incidence of IKBKG and IKBKGP recombination. Because these two genes are in opposite position, recombination after DNA loop back is likely to occur in somatic cells. The investigators will transform lymphocytes containing IKBKGP mutation, and culture them continuously. IKBKG mutation will be check intermittently and the incidence can be estimated. The third aim is to find a treatment. The investigators will test the read-through drug gentamycin and PTC2124 for nonsense mutation. Either fibroblast or Epstein-Barr virus (EBV) - transformed lymphoblasts will be tested. The investigators hope this study with not only increases our understand to IP, and also improves the investigators' knowledge toward genetic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed to have Incontinentia Pigmenti

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Incontinentia Pigmenti
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Mutation analysis result | 1 year
  Mutation analysis result

CONTACTS AND LOCATIONS:
Overall Officials: NiChung Lee, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan